CLINICAL TRIAL: NCT05886348
Title: The Evaluation of Safety and Myopia Progression Control Using Novel Spectacle Lens
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HOYA Lens Thailand LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DG2-3A
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Model-A Novel Spectacle lens (Experimental)
  Interventions: Device: Model-A Novel spectacle lens
- Model-B Novel Spectacle lens (Experimental)
  Interventions: Device: Model-B Novel spectacle lens
- Single Vision Spectacle lens (Other)
  Interventions: Device: Single vision spectacle lens

INTERVENTIONS:
Device: Model-A Novel spectacle lens — Model-A Novel spectacle lenses will be given to 1 arm to wear for 36 months
  Arms: Model-A Novel Spectacle lens
Device: Model-B Novel spectacle lens — Model-B Novel spectacle lenses will be given to 1 arm to wear for 36 months
  Arms: Model-B Novel Spectacle lens
Device: Single vision spectacle lens — Single Vision Spectacle lenses will be given to 1 arm to wear for 36 months
  Arms: Single Vision Spectacle lens

SUMMARY:
The goal of this clinical trial is to test Novel spectacle lenses in myopic children. The main question it aims to answer are: safety and efficacy of the lenses. Participants will be asked to wear spectacles and participate in eye exams and questionnaires. Researchers will compare Novel spectacle lenses and general single vision spectacle lenses to see if the Novel spectacle lenses correct myopic ametropia, slow the progression of myopia and axial elongation.

DETAILED DESCRIPTION:
This is a 3-year prospective, multicenter, randomized, and single-masked*, parallel-group controlled clinical study. The purpose of this study is to evaluate the safety and efficacy of wearing Novel spectacle lenses to correct myopic ametropia, slow the progression of myopia and axial elongation in myopic children as compared to the use of single vision spectacles lenses.

The treatment arms are:

* Model A Novel spectacle lens
* Model B Novel spectacle lens
* Single vision spectacle lens

Single-masked:

The investigator responsible for conducting ocular data measurements related to the primary and secondary endpoints will be masked. The participants will not be informed the treatment arm during the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Participant and parent (or guardian) are able and willing to provide consent
2. Participant and parent (or guardian) ensure to attend required study visits and adhere to participant requirements
3. Parent or guardian understands and accepts random allocation of grouping, and that participant and parent (or guardian) will not be told which group participant is allocated to
4. Participant willing to wear the study spectacles lens for a minimum of 12 hours per day for the duration of the study
5. Age at time of parent or guardian consent and participant assent: 7 - 13 years old
6. Spherical equivalent cycloplegic autorefraction: -1.00 to -7.00 D in each eye.
7. Cycloplegic autorefraction astigmatism of 1.50 D or less in each eye
8. Cycloplegic autorefraction anisometropia of 1.50 D or less
9. Monocular best corrected distance visual acuity (BCDVA) equal to or better than logMAR 0.10 in each eye.

Exclusion Criteria:

1. Participant is allergy to fluorescein, benoxinate, proparacaine, tropicamide or cyclopentolate eye drops
2. Any ocular and systemic abnormalities might be expected to affect visual functions or refractive development
3. (a) Have received treatment of myopic control pharmaceutical medication (e.g., atropine) or light fundus illuminance therapy (e.g., repeated red light therapy) within 6 months prior to entry into this study. (b) Have received treatment of myopia control such as contact lenses, orthokeratology lenses etc., progressive addition lenses, bifocal lenses, within 3 months. (c) Have received treatment of myopia control such as defocus spectacle lenses (difference between both eye's non-cycloplegic autorefraction and lens-meter results of the respective lenses are equal or less than 0.50 D SER) etc. within one month prior to entry into this study.
4. Participant with clinically significant strabismus (including intermittent tropia)
5. Medical history of binocular vision abnormalities
6. Participant with amblyopia
7. Participation in a clinical trial within 30 days prior to entry into this study or during participation
8. Previous intraocular surgery
9. Participant who, in the judgment of the Investigator, presence of any emotional, physiologic, or anatomical condition which may preclude participation in this study or provide an inappropriate landscape for the intended study treatment.
10. Any medical treatment or medication which might have an influence on vision or interfere with study assessments
11. Pathological myopia (myopia that leads to structural changes in the posterior segment of the eye including posterior staphyloma, myopic maculopathy, and high myopia-associated optic neuropathy)

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 249 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Axial length | 24 months
  The difference of Axial length changes over 24 months between treatment groups in low and moderate myopia (-1.00 D to -5.00 D) participants.
Spherical equivalent cycloplegic autorefraction | 24 months
  The difference of spherical equivalent cycloplegic autorefraction changes over 24 months between treatment groups in low and moderate myopia (-1.00 D to -5.00 D) participants

SECONDARY OUTCOMES:
Axial length | 36 months
Spherical equivalent cycloplegic autorefraction | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: William Zhou, MD, Study Chair — HOYA Lens Thailand LTD.
Locations (5):
- China (5):
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - Guangzhou Aier Eye Hospital, Guangzhou
  - Eye and ENT Hospital of Fudan University, Shanghai
  - Shengyang He Eye Specialist Hospital, Shengyang
  - Tianjin Medical University Eye Hospital, Tianjin